CLINICAL TRIAL: NCT05349643
Title: A Phase 2, Open-Label, Adaptive, Dose-Ranging Study With Long-Term Extension to Evaluate the Safety, Tolerability, Efficacy, and Pharmacokinetics of Intra Articular AMB-05X Injections in Subjects With Tenosynovial Giant Cell Tumor
Brief Title: A Study to Evaluate Safety and Efficacy of AMB-05X Injections in Subjects With TGCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AmMax Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMB-051-07
Record Dates: First submitted 2022-04-22; First posted 2022-04-27 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Pigmented Villonodular Synovitis; TGCT; Tenosynovial Giant Cell Tumor
Keywords: Pigmented Villonodular Synovitis; Tenosynovial Giant Cell Tumor; TGCT; PVNS
MeSH Terms: conditions — Synovitis, Pigmented Villonodular; Giant Cell Tumor of Tendon Sheath

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMB-05X (Experimental): Subjects will receive an injection of AMB-05X once every 4 weeks for 24 weeks (for 6 treatments total). Based on ongoing review of the available safety, PK, PD, and efficacy data, the Sponsor may either increase or decrease the dose.
  Interventions: Biological: AMB-05X

INTERVENTIONS:
Biological: AMB-05X — A fully human monoclonal immunoglobulin (IgG2) directed against c-fms

SUMMARY:
AMB-051-07 is an open-label, adaptive, dose-ranging study with long-term extension in adults with tenosynovial giant cell tumor

DETAILED DESCRIPTION:
AMB-051-07 is an open-label, adaptive, dose-ranging study with long-term extension which will enroll up to 48 adult subjects with tenosynovial giant cell tumor for intra-articular doses over a 24-week dosing period (Part 1) with a Part 2 open-label extension of 6 treatment and/or observational cycles of 12 weeks each followed by 12 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subject ≥ 18 years
2. TGCT with only 1 joint involvement
3. Symptomatic Measurable disease of at least 1 cm based on RECIST v1.1
4. Stable prescription of analgesic regimen
5. Agrees to follow contraception guidelines
6. Women of childbearing potential must have a negative pregnancy test
7. Adequate hematologic, hepatic, and renal function

Exclusion Criteria:

1. Prior investigational drug use within 4 weeks or 5 half-lives of Baseline
2. Previous use of therapeutics targeting CSF1 or CSF1R or oral tyrosine kinase inhibitors within 3 months prior to Baseline
3. History of extensive or reconstructive surgery on the affected joint
4. Active cancer (either currently or within 3 mo before Baseline) that requires/required therapy (e.g., surgery, chemotherapy, or radiation therapy)
5. Metastatic or malignant transformation of TGCT
6. Hepatitis C virus (HCV) or hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
7. Known active tuberculosis
8. Significant concomitant arthropathy in the affected joint, serious illness, uncontrolled infection, or a medical or psychiatric history
9. Women who are breastfeeding
10. A screening Fridericia-corrected QT interval (QTcF) ≥ 470 ms
11. MRI contraindications (e.g., pacemaker, loose metallic implants)
12. History of hypersensitivity to any ingredient of the study drug
13. History of drug or alcohol abuse within 3 months before baseline
14. Any other severe acute or chronic medical or psychiatric condition or clinically significant laboratory abnormality that may increase the risk associated with study participation/treatment or interfere with interpretation of study results and, in the Investigator's opinion, make the subject inappropriate for this study
15. Subjects who, in the Investigator's opinion, should not participate in the study for any reason, including if there is a question about their ability to comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate - Part 1 | Part 1 Week 24
  Proportion of subjects who achieve an OR (objective response rate [ORR]) by central radiology review per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Treatment-emergent adverse events | Part 1 Week 24 and Part 2 Week 72
  Frequency and severity of reported treatment-emergent adverse events

SECONDARY OUTCOMES:
Objective Response Rate | Part 2 Week 72
  Proportion of subjects who achieve an OR (objective response rate [ORR]) by central radiology review per modified Response Evaluation Criteria in Solid Tumors
Objective Response Rate (AMB-051-01 subjects) | Part 2 Week 72
  Proportion of re-treated subjects who achieve an OR (objective response rate [ORR]) by central radiology review per modified Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
Objective Response Rate (ORR) per modified Response Evaluation Criteria in Solid Tumors Version 1.1 | Part 1 Week 24
  Proportion of subjects who achieve an overall response (OR) per modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Objective Response Rate (ORR) per modified Response Evaluation Criteria in Solid Tumors Version 1.1 | Part 2 Week 72
  Proportion of subjects who achieve an overall response (OR) per modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Tumor response based on tumor volume score (TVS) | Part 1 Week 24
  Proportion of subjects who achieve an overall tumor response (OR) per the tumor volume score
Tumor response based on tumor volume score (TVS) | Part 2 Week 72
  Proportion of subjects who achieve an overall tumor response (OR) per the tumor volume score
Duration of Response by Response Evaluation Criteria in Solid Tumors | Part 1 Week 24
  Median duration of response per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Duration of Response by Response Evaluation Criteria in Solid Tumors v1.1 | Part 2 Week 72
  Median duration of response per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Duration of Response by Modified Response Evaluation Criteria in Solid Tumors | Part 1 Week 24
  Median duration of response per modified Response Evaluation Criteria in Solid Tumors (modified RECIST)
Duration of Response by Modified Response Evaluation Criteria in Solid Tumors | Part 2 Week 72
  Median duration of response per modified Response Evaluation Criteria in Solid Tumors (modified RECIST)
Duration of Response by tumor volume score | Part 1 Week 24
  Median duration of response per tumor volume score (TVS)
Duration of Response by tumor volume score | Part 2 Week 72
  Median duration of response per tumor volume score (TVS)
Time to Response by Response Evaluation Criteria in Solid Tumors | Part 1 Week 24
  Time to response (TTR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Time to Response by Response Evaluation Criteria in Solid Tumors | Part 2 Week 72
  Time to response (TTR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Time to Response by Modified Response Evaluation Criteria in Solid Tumors | Part 1 week 24
  Time to response (TTR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Time to Response by Modified Response Evaluation Criteria in Solid Tumors | Part 2 Week 72
  Time to response (TTR) per modified Response Evaluation Criteria in Solid Tumors (modified RECIST)
Time to Response per tumor volume score | Part 1 Week 24
  Time to response (TTR) per tumor volume score (TVS)
Time to Response per tumor volume score | Part 2 Week 72
  Time to response (TTR) per tumor volume score (TVS)
Mean change from Baseline in joint range of motion (ROM) | Part 1 Week 24
  Mean change in joint range of motion (ROM) will be assessed by qualified assessors. Measurements will be recorded in degrees. At baseline, the plane of movement with the smallest (worst) relative value will be identified; only this plane will be used for evaluating change in ROM subsequently.
Mean change from Baseline in joint range of motion (ROM) | Part 2 Week 72
  Mean change in joint range of motion (ROM) will be assessed by qualified assessors. Measurements will be recorded in degrees. At baseline, the plane of movement with the smallest (worst) relative value will be identified; only this plane will be used for evaluating change in ROM subsequently.
Mean change from Baseline in the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function score | Part 1 Week 24
  The Patient-Reported Outcomes Measurement Information System (PROMIS) is a 10-question patient reported outcome instrument used to assess physical functioning based on use of the upper extremities (dexterity), lower extremities (walking or mobility), and central regions (neck, back) and on instrumental activities of daily living. Five questions address the degree to which subject's health limits activities; subjects select responses ranging from 1-cannot do to 5 - not at all. Five additional questions address the degree to which the subject is able to perform certain physical activities, and subjects select a response to each question that ranges from 1 ("cannot do") to 5 ("without any difficulty"). Raw scores are summarized, score range is 10 to 50.
Mean change from Baseline in the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function score | Part 2 Week 72
  The Patient-Reported Outcomes Measurement Information System (PROMIS) is a 10-question patient reported outcome instrument used to assess physical functioning based on use of the upper extremities (dexterity), lower extremities (walking or mobility), and central regions (neck, back) and on instrumental activities of daily living. Five questions address the degree to which subject's health limits activities; subjects select responses ranging from 1-cannot do to 5 - not at all. Five additional questions address the degree to which the subject is able to perform certain physical activities, and subjects select a response to each question that ranges from 1 ("cannot do") to 5 ("without any difficulty"). Raw scores are summarized, score range is 10 to 50.
Mean change from Baseline in Worst Stiffness Numeric Rating Scale score | Part 1 Week 24
  The Worst Stiffness Numeric Rating Scale (NRS) is a 1-item, self-administered questionnaire assessing the "worst" stiffness within the last 24 hours. The NRS for this item ranges from 0 (no stiffness) to 10 (stiffness as bad as you can imagine). Higher scores indicate worst stiffness.
Mean change from Baseline in Worst Stiffness Numeric Rating Scale score | Part 2 Week 72
  The Worst Stiffness Numeric Rating Scale (NRS) is a 1-item, self-administered questionnaire assessing the "worst" stiffness within the last 24 hours. The NRS for this item ranges from 0 (no stiffness) to 10 (stiffness as bad as you can imagine). Higher scores indicate worst stiffness.
Mean change from Baseline in the Brief Pain Inventory (BPI) score | Part 1 Week 24
  Brief Pain Inventory (BPI) Short Form is a self-administered questionnaire used to evaluate the severity of a subject's pain and the impact of this pain on the subject's daily functioning. The subject is asked to rate their worst, least, average, and current pain intensity, list current treatments and their perceived effectiveness, and rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a scale from 0 ="no pain" to 10= "pain as bad as you can imagine".
Mean change from Baseline in the Brief Pain Inventory (BPI) score | Part 2 Week 72
  Brief Pain Inventory (BPI) Short Form is a self-administered questionnaire used to evaluate the severity of a subject's pain and the impact of this pain on the subject's daily functioning. The subject is asked to rate their worst, least, average, and current pain intensity, list current treatments and their perceived effectiveness, and rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a scale from 0 ="no pain" to 10="pain as bad as you can imagine".
Decrease of at least 30% in mean Brief Pain Inventory (BPI) from Baseline | Part 1 Week 24
  Brief Pain Inventory (BPI) Short Form is a self-administered questionnaire used to evaluate the severity of a subject's pain and the impact of this pain on the subject's daily functioning. The subject is asked to rate their worst, least, average, and current pain intensity, list current treatments and their perceived effectiveness, and rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a scale from 0 ="no pain" to 10="pain as bad as you can imagine".
Decrease of at least 30% in mean Brief Pain Inventory (BPI) from Baseline | Part 2 Week 72
  Brief Pain Inventory (BPI) Short Form is a self-administered questionnaire used to evaluate the severity of a subject's pain and the impact of this pain on the subject's daily functioning. The subject is asked to rate their worst, least, average, and current pain intensity, list current treatments and their perceived effectiveness, and rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a scale from 0 ="no pain" to 10="pain as bad as you can imagine".
Mean change from Baseline in Patient-Reported Outcomes Measurement Information System Pain Interference score | Part 1 Week 24
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v1.1 Pain Interference Short Form 8a, is an 8 question instrument used to evaluate how much a subject's pain interferes with daily functioning. Subjects rate the degree to which pain interfered with their daily activity over the past 7 days on a scale of 1 to 5 (ranging from 1, "Not at all," to 5, "Very much"). Higher scores indicate greater pain interference.
Mean change from Baseline in Patient-Reported Outcomes Measurement Information System Pain Interference score | Part 2 Week 72
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v1.1 Pain Interference Short Form 8a, is an 8 question instrument used to evaluate how much a subject's pain interferes with daily functioning. Subjects rate the degree to which pain interfered with their daily activity over the past 7 days on a scale of 1 to 5 (ranging from 1, "Not at all," to 5, "Very much"). Higher scores indicate greater pain interference.
Mean change from Baseline in Patient Global Impression of Change in Physical Functioning for capacity to perform everyday tasks | Part 1 Week 24
  The Patient Global Impression of Change (PGIC), also known as Subject Global Impression. For this study, subjects will rate how much their tenosynovial giant cell tumor (TGCT) has restricted their ability to perform everyday tasks, using the following scales that are based on the PGIC: PGIC Physical Functioning scale (ranging from 1 "Not at all," to 5 "Extremely" and rate their change in stiffness using the PGIC Stiffness scale (ranging from 1 "Very much improved" to 7 "Very much worse". Higher scores indicate greater restrictions.
Mean change from Baseline in Patient Global Impression of Change in Physical Functioning for capacity to perform everyday tasks | Part 2 Week 72
  The Patient Global Impression of Change (PGIC), also known as Subject Global Impression. For this study, subjects will rate how much their tenosynovial giant cell tumor (TGCT) has restricted their ability to perform everyday tasks, using the following scales that are based on the PGIC: PGIC Physical Functioning scale (ranging from 1, "Not at all," to 5, "Extremely" and rate their change in stiffness using the PGIC Stiffness scale (ranging from 1 "Very much improved" to 7 "Very much worse". Higher scores indicate greater restrictions.
Mean change from Baseline in Patient Global Impression of Change in tenosynovial giant cell tumor-related stiffness score | Part 1 Week 24
  The Patient Global Impression of Change (PGIC), also known as Subject Global Impression. For this study, subjects will rate how much their tenosynovial giant cell tumor (TGCT) has restricted their ability to perform everyday tasks, using the PGIC to rate their change in stiffness using the PGIC Stiffness scale, ranging from 1, "Very much improved" to 7, "Very much worse". Higher scores indicate greater TGCT-related levels of stiffness.
Mean change from Baseline in Patient Global Impression of Change in tenosynovial giant cell tumor-related stiffness score | Part 2 Week 72
  The Patient Global Impression of Change (PGIC), also known as Subject Global Impression. For this study, subjects will rate how much their TGCT has restricted their ability to perform everyday tasks, using the PGIC to rate their change in stiffness using the PGIC Stiffness scale, ranging from 1, "Very much improved" to 7, "Very much worse". Higher scores indicate greater TGCT-related levels of stiffness.
Mean change from Baseline in Worst Pain Numeric Rating Scale score | Part 1 Week 24
  The Worst Pain Numeric Rating Scale (NRS) is an item in the Brief Pain Inventory (BPI) that assesses a subject's "worst" pain in the last 24 hours. The 11-point NRS for this item ranges from 0 ("no pain") to 10 ("pain as bad as you can imagine"). Higher scores indicate greater levels of pain.
Mean change from Baseline in Worst Pain Numeric Rating Scale score | Part 2 Week 72
  The Worst Pain Numeric Rating Scale (NRS) is an item in the Brief Pain Inventory (BPI) that assesses a subject's "worst" pain in the last 24 hours. The 11-point NRS for this item ranges from 0 ("no pain") to 10 ("pain as bad as you can imagine"). Higher scores indicate greater levels of pain.
EuroQol 5 Dimension 5 Level Health Assessment | Part 1 Week 24
  EuroQol 5 Dimension 5 Level (EQ-5D-5L) is a widely used quality of life instrument that includes questions in each of 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The choices include 5 levels of severity for each domain followed by a general health visual analogue scale (VAS). This instrument is a self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking that ranges from "no problems" through "extreme problems". Higher scores indicate a lower quality of life.
EuroQol 5 Dimension 5 Level Health Assessment | Part 2 Week 72
  EuroQol 5 Dimension 5 Level (EQ-5D-5L) is a widely used quality of life instrument that includes questions in each of 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The choices include 5 levels of severity for each domain followed by a general health visual analogue scale (VAS). This instrument is a self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking that ranges from "no problems" through "extreme problems". Higher scores indicate a lower quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Nguyen, MD, Study Chair — AmMax Bio
Locations (6):
- United States (3):
  - AmMax Bio, Clinical Site, Sacramento, California
  - AmMax Bio, Clinical Site, Miami, Florida
  - AmMax Bio, Clinical Site, Houston, Texas
- Australia (2):
  - AmMax Bio, Clinical Site, Camperdown
  - AmMax Bio, Clinical Site, Woolloongabba
- AmMax Bio, Clinical Site, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No